CLINICAL TRIAL: NCT06487390
Title: PrEP Pro: Adapting a Multi-component Intervention to Train and Support Providers to Promote PrEP for Adolescent Girls and Young Women in the Deep South
Brief Title: Multi-component Intervention to Train Providers to Promote PrEP for Girls and Women in the Deep South
Acronym: PrEP Pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lynn T. Matthews, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300008567; R34MH128044-01 (NIH)
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: PrEP; HIV; HIV prevention; Adolescents; Young adults; Family Medicine; Residents; Physician Trainees; Training intervention; Sexual history; Sexual Health; Sexually Transmitted Infections
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resident Trainees (Experimental): Family medicine resident trainees who receive the PrEP Pro training intervention
  Interventions: Behavioral: PrEP Pro training intervention

INTERVENTIONS:
Behavioral: PrEP Pro training intervention — Training intervention adapted from evidence-based HIV epidemiology, sexual history taking, and PrEP prescription curricula.

SUMMARY:
The goal of this study is to adapt evidence-based curriculum on HIV epidemiology and PrEP prescription to train family medicine physician trainees to take a thorough sexual history and discuss HIV/STI prevention and PrEP options with adolescent patients in Alabama. The primary outcomes of the study are:

* Feasibility of the PrEP Pro training intervention
* Acceptability of the PrEP Pro training intervention

Secondary outcomes include:

* Behavioral changes in sexual history taking performed by physician trainees
* PrEP knowledge and prescribing practices
* HIV and STI screening practices

Participants will receive training on sexual history taking and HIV prevention options, including PrEP prescription and management. They will complete a pre-training survey (enrollment) and post-training survey (6 months post enrollment) to understand differences in knowledge and practice before and after receiving the training intervention. The post training survey will also assess acceptability and feasibility of the intervention. A subset of participants will complete qualitative in-depth interviews to further discuss their experiences with the program and suggestions for future adaptations.

ELIGIBILITY:
Inclusion Criteria:

1. licensed HCP (MD, DO) trainee
2. providing medical care to AGYW in AL
3. working in a clinic setting where at least 20% of the population is Black
4. able/willing to provide informed consent

Exclusion Criteria:

(a) unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Latesha E. Elopre, MD, MSPH, Principal Investigator — University of Alabama at Birmingham; Lynn T Matthews, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- See also: PrEP Pro Protocol Paper — https://pubmed.ncbi.nlm.nih.gov/36943364/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Alabama study involved 4 family medicine residency programs across 5 clinical sites. We contacted 10 of 11 known programs (as of 2023); 4 agreed to participate. Three others had participated in earlier phases but lacked sufficient resident turnover to participate further. Partner sites delivered the intervention training, and trained residents could opt into study participation by completing baseline/exit surveys or in-depth interviews.
Groups:
- PrEP Pro Participants (Pilot Test): Family medicine resident trainees and PrEP Champions (residents and/or faculty) who received the PrEP Pro training intervention during the pilot test
Period: Overall Study
Arm/Group | PrEP Pro Participants (Pilot Test)
Started | 46
Completed | 32
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | PrEP Pro Participants (Pilot Test)
Number analyzed (Participants) | 46
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/gender as reported by participants
  Participants
    Sex/gender: Female | 19
    Sex/gender: Male | 26
    Sex/gender: Gender nonconforming | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity as reported by participants
  Participants
    Hispanic or Latino | 5
    Not Hispanic or Latino | 41
    Unknown or Not Reported | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Age in years as reported by participants
  years | 29 [28 to 33.75]
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — 8 race categories including missing and more than one race; categories are mutually exclusive -- those who reported more than one race were categorized as "more than one race" rather the individually selected races
  Participants
    Race: American Indian or Alaskan Native | 0
    Race: Asian | 6
    Race: Native Hawaiian or Other Pacific Islander | 0
    Race: Black or African American | 2
    Race: White | 26
    Race: More than one race | 2
    Race: Unknown/missing | 3
    Race: Middle Eastern or North African | 7
HIV Epidemiology knowledge assessment [Number; unit: Percentage of Participants] — Measured by baseline and 6-month (pre- and post-training) surveys; scores range from 0-100% based on the percentage of participants who answered all five questions related to HIV epidemiology correctly; higher percentages indicate that more participants knew the correct answer to all 5 HIV epidemiology questions. Population: 46 pilot test participants completed the baseline questionnaire.
  Percentage of Participants | 17.39
Sexual History Taking Practices [Median (Inter-Quartile Range); unit: Scores of a scale] — Measured by baseline survey. Sexual history taking knowledge, attitudes, and beliefs. 23 questions split into four subscales on 3-point Likert scale; each subscale score is the mean of the scores from the questions in the scale.
  Subscales: Attitudes (4 items), Skills (14), Barriers (2), Training (3). Strongly agree/Somewhat agree = 3, Neither agree nor disagree = 2, Strongly disagree/Somewhat disagree = 1 Higher score on 1-3 range indicates more positive attitude towards sexual history assessment, higher skill, more barriers, and better training. Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire. Baseline and Exit questionnaires were scored looking only at participants who completed both.
  Scores of a scale
    Attitudes: number analyzed (Participants) | 32
    Attitudes | 2.5 [2.5 to 2.8]
    Skills: number analyzed (Participants) | 32
    Skills | 2.9 [2.8 to 3.0]
    Barriers: number analyzed (Participants) | 32
    Barriers | 3.0 [2.0 to 3.0]
    Training: number analyzed (Participants) | 32
    Training | 2.7 [2.3 to 2.8]
PrEP Knowledge, Willingness to Prescribe, Prescribing Practices [Mean (Inter-Quartile Range); unit: scores on a scale] — measured by baseline and 6-month (pre- and post-training) surveys, qualitative interviews, EMR data.
  The score ranges for each subscale varied (PrEP knowledge=0-20, attitudes=0-28, and beliefs=0-8), with high values on each subscale representing good knowledge or positive attitudes toward PrEP, respectively. Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire. Baseline and Exit questionnaires were scored looking only at participants who completed both.
  scores on a scale
    Baseline PrEP knowledge (score 0-20): number analyzed (Participants) | 32
    Baseline PrEP knowledge (score 0-20) | 9.5 [4 to 14]
    Baseline PrEP attitudes (score 0-28): number analyzed (Participants) | 32
    Baseline PrEP attitudes (score 0-28) | 24 [21 to 26]
    Baseline PrEP beliefs (score 0-8): number analyzed (Participants) | 32
    Baseline PrEP beliefs (score 0-8) | 6 [5 to 8]
STI screening practices [Number; unit: Percent of Participants] — Percent of participants who reported assessing sexual history and/or testing clients for STIs in the past week at least some of the time, by group (AGYW/ABYM).
  "At least some of the time" = answering "some, many, most, or all" (vs "none") to questions formatted like: Among the [AGYW/ABYM] seen last week, for about how many did you [assess sex Hx/test for STIs]?
  measured by BL and 6-month surveys, IDIs, EMR data; BL=baseline; AGYW=adolescent girls and young women (ages 14-24); ABYM=adolescent boys and young men (ages 14-24); sex Hx=assessed for sexual history; past wk=past 7 days Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire. Baseline and Exit questionnaires were scored looking only at participants who completed both.
  Percent of Participants
    BL AGYW sex Hx past wk: number analyzed (Participants) | 32
    BL AGYW sex Hx past wk | 78.13
    BL AGYW tested for STI past wk: number analyzed (Participants) | 32
    BL AGYW tested for STI past wk | 53.13
    BL ABYM sex Hx past wk: number analyzed (Participants) | 32
    BL ABYM sex Hx past wk | 78.13
    BL ABYM tested for STI past wk: number analyzed (Participants) | 32
    BL ABYM tested for STI past wk | 28.13
HIV screening practices [Number; unit: Percentage of Participants] — Percent of participants (providers) who reported they tested clients for HIV in the past week at least some of the time, by group (AGYW/ABYM).
  "At least some of the time" = answering "some, many, most, or all" (vs "none") to questions formatted like: Among the [AGYW/ABYM] seen last week, for about how many did you [test for HIV]?
  measured by BL and 6-month surveys, IDIs, EMR data; BL=baseline; AGYW=adolescent girls and young women (ages 14-24); ABYM=adolescent boys and young men (ages 14-24); sex Hx=assessed for sexual history; past wk=past 7 days Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire. Baseline and Exit questionnaires were scored looking only at participants who completed both.
  Percentage of Participants
    BL AGYW tested for HIV past wk: number analyzed (Participants) | 32
    BL AGYW tested for HIV past wk | 28.13
    BL ABYM tested for HIV past wk: number analyzed (Participants) | 32
    BL ABYM tested for HIV past wk | 21.88

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Intervention Implementation
Description: Feasibility of Intervention: 4 items, 5-point Likert scale, scale values range from 1-5 with higher score meaning more feasible to implement
Time Frame: 6 months
Population: Due to a technical error in the questionnaire software, among the 32 exit questionnaire participants, 17 completed the acceptability, feasibility, and appropriateness measures.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 17
Scores on a scale | 4.28 (0.42)

2. Primary Outcome: Acceptability
Description: Acceptability of Intervention: 4 items, 5-point Likert scale, scale values range from 1-5 with higher score meaning the intervention is more acceptable to participants
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- PrEP Pro participants (Pilot Test): Family medicine resident trainees and PrEP Champions (residents and/or faculty) who received the PrEP Pro training intervention during the pilot test phase
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 17
Scores on a scale | 4.31 (0.53)

3. Secondary Outcome: HIV Epidemiology Knowledge Assessment
Description: Measured by baseline and 6-month (pre- and post-training) surveys; scores range from 0-100% based on the percentage of participants who answered all five questions related to HIV epidemiology correctly; higher percentages indicate that more participants knew the correct answer to all 5 HIV epidemiology questions.
Time Frame: 6 months
Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire.
Measure: Number; unit: Percentage of Participants
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 32
Percentage of Participants | 18.75

4. Secondary Outcome: Sexual History Taking Practices
Description: Measured by baseline survey. Sexual history taking knowledge, attitudes, and beliefs. 23 questions split into four subscales on 3-point Likert scale; each subscale score is the mean of the scores from the questions in the scale.
  Subscales: Attitudes (4 items), Skills (14), Barriers (2), Training (3). Strongly agree/Somewhat agree = 3, Neither agree nor disagree = 2, Strongly disagree/Somewhat disagree = 1 Higher score on 1-3 range indicates more positive attitude towards sexual history assessment, higher skill, more barriers, and better training.
Time Frame: 6 months
Population: N=32 out of 46 pilot test participants chose to take the exit questionnaire. Baseline and Exit questionnaires were scored looking only at participants who completed both.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 32
scores on a scale
  Attitudes | 2.5 [2.5 to 2.8]
  Skills | 3.0 [2.9 to 3.0]
  Barriers | 3 [2.5 to 3.0]
  Training | 2.7 [2.3 to 3.0]

5. Secondary Outcome: PrEP Knowledge, Willingness to Prescribe, Prescribing Practices
Description: measured by baseline and 6-month (pre- and post-training) surveys, qualitative interviews, EMR data.
  The score ranges for each subscale varied (PrEP knowledge=0-20, attitudes=0-28, and beliefs=0-8), with high values on each subscale representing good knowledge or positive attitudes toward PrEP, respectively.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Inter-Quartile Range); unit: scores on a scale
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 32
scores on a scale
  Exit Questionnaire (EQ) PrEP knowledge (score 0-20) | 16 [13 to 19]
  EQ PrEP attitudes (score 0-28) | 26 [23 to 28]
  EQ PrEP beliefs (score 0-8) | 6 [5 to 7]

6. Secondary Outcome: STI Screening Practices
Description: Percent of participants (providers) who reported they assessed sexual history and/or tested clients for STIs in the past week at least some of the time, by group (AGYW/ABYM).
  "At least some of the time" = answering "some, many, most, or all" (vs "none") to questions formatted like: Among the [AGYW/ABYM] seen last week, for about how many did you [assess sex Hx/test for STIs]?
  measured by BL and 6-month surveys, IDIs, EMR data; BL=baseline; AGYW=adolescent girls and young women (ages 14-24); ABYM=adolescent boys and young men (ages 14-24); sex Hx=assessed for sexual history; past wk=past 7 days
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: Percent of Participants
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 32
Percent of Participants
  Exit AGYW assessed sexual history in the past week | 90.63
  Exit AGYW tested for STI in the past week | 56.25
  Exit Adolescent boys/young men (ABYM) assessed sexual history in the past week | 71.88
  Exit ABYM tested for STI in the past week | 34.38

7. Secondary Outcome: HIV Screening Practices
Description: Percent of participants (providers) who reported they tested clients for HIV in the past week at least some of the time, by group (AGYW/ABYM).
  "At least some of the time" = answering "some, many, most, or all" (vs "none") to questions formatted like: Among the [AGYW/ABYM] seen last week, for about how many did you [test for HIV]?
  measured by BL and 6-month surveys, IDIs, EMR data; BL=baseline; AGYW=adolescent girls and young women (ages 14-24); ABYM=adolescent boys and young men (ages 14-24); sex Hx=assessed for sexual history; past wk=past 7 days
Time Frame: 6 months
Population: as for outcome 4
Measure: Number; unit: Percent of Participants
Arm/Group | PrEP Pro participants (Pilot Test)
Number analyzed (Participants) | 32
Percent of Participants
  Exit AGYW tested for HIV in the past week | 40.63
  Exit ABYM tested for HIV in the past week | 28.13

ADVERSE EVENTS:
Time Frame: from enrollment until the end of the trial period (6 month pilot test)
Arm/Group | PrEP Pro Participants (Pilot Test)
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

LIMITATIONS AND CAVEATS:
This study is limited by small sample size, short follow-up, and sampling bias from clinics that opted in. Effectiveness in improving PrEP prescribing could not be assessed. The intervention did not address provider stigma or restrictive state laws.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT06487390/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT06487390/ICF_001.pdf